CLINICAL TRIAL: NCT04069884
Title: RecurIndex Guided Avoidance of Regional Nodal Irradiation for Node Positive Breast Cancer
Acronym: RIGAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaobo Huang, Head of Breast Radiotherapy, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIGAIN
Record Dates: First submitted 2019-08-19; First posted 2019-08-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Radiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Clinical low-risk, RecurIndex high-risk) (Experimental): Regional nodal irradiation (RNI) was given along with whole breast irradiation (WBI) or Chest wall irradiation (CWI) for breast-conserving patients and total mastectomy patients, respectively.
  Interventions: Radiation: regional nodal irradiation; Radiation: WBI; Radiation: chestwall XRT
- Arm II (Clinical low-risk, RecurIndex high-risk) (Active Comparator): No Regional nodal irradiation (RNI) , whole breast irradiation (WBI) for breast-conserving patients and No Chest wall irradiation (CWI) for total mastectomy patients.
  Interventions: Radiation: WBI

INTERVENTIONS:
Radiation: regional nodal irradiation — external-beam radiotherapy (XRT)
  Arms: Arm I (Clinical low-risk, RecurIndex high-risk)
Radiation: WBI — Whole Breast Irradiation
Radiation: chestwall XRT — chestwall irradiation
  Arms: Arm I (Clinical low-risk, RecurIndex high-risk)

SUMMARY:
The purpose of this study is to validate whether clinically low-risk, and RecurIndex high-risk N1 patients receiving regional lymph node radiotherapy can further improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, ≤ 70 years old.
* Eastern Cooperative Oncology Group (ECOG) ≤ 2.
* Postoperative pathology is clearly diagnosed as invasive breast cancer.
* Meet the clinical definition of low risk: ①Axillary lymph node micrometastasis (N1mic) or ②N1 patients who meet the following conditions at the same time, a）Age ≥ 40 years old, b）Vascular tumor thrombus (LVI) negative or allow few positive LVI (excluding extensive or massive LVI), c）Three subtypes are allowed (Lumina A, Lumina B/HER2 negative, Lumina B/HER2 positive) , namely ER positive (ER ≥ 1%), HER2 negative (HER2 expression negative or + by IHC, or 2+ but negative by FISH) or ER positive (ER ≥ 1%), HER2 positive (3+ by IHC, or 2+ but positive by FISH).
* Postoperative pathological diagnosis of axillary lymph node status is any of the following: a. Sentinel lymph node biopsy or axillary lymph node dissection for micrometastasis (N1mic), b. Sentinel lymph node biopsy for 1-2 lymph node macrometastasis (N1sln), c. Sentinel lymph node biopsy + axillary lymph node dissection or simple axillary lymph node dissection for 1-3 lymph node metastasis (N1).
* The primary tumor and breast undergo breast-conserving surgery or total resection ± breast reconstruction (autologous/prosthetic).
* There must be adequate systemic examination (such as chest X-ray, B-ultrasound, CT, etc.) within 3 months before randomization of radiotherapy to confirm that there is no distant metastasis.
* No contralateral breast cancer must be confirmed by molybdenum target and/or MRI within 12 months before randomization of radiotherapy.
* At least 4 courses of adjuvant chemotherapy with anthracycline or taxane should be completed after surgery. If patients with HR positive, HER2 negative tumor underwent Multigene Assays, with low risk scores, omitting chemotherapy is permitted.
* Radiotherapy must be performed sequentially after the completion of adjuvant chemotherapy, starting no later than 8 weeks after the end of chemotherapy.
* The patient must have sufficient primary fresh frozen specimens or post-paraffin tissue sections for RecurIndex testing.
* No previous history of malignant tumors, except for basal cell carcinoma of the skin.
* Signed an informed consent form.

Exclusion Criteria:

* Postoperative radiotherapy was confirmed as T3-4, N0, N2-3, M1 lesion staging before enrollment.
* Receive any new adjuvant therapy before surgery, including chemotherapy, endocrine therapy, targeted therapy or radiation therapy.
* Patients who underwent total mastectomy and only sentinel lymph node biopsy.
* Have a history of contralateral breast cancer.
* History of chest radiotherapy.
* combined with severe heart, lung, liver, kidney, hematopoietic, neurological diseases, and mental illness.
* History of autoimmune diseases such as scleroderma or active lupus erythematosus.
* pregnant and lactating patients.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2029-08-20 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival (IDFS) | 5 years
  defined as the time between randomization and either local recur, distant metastases or death occurred

SECONDARY OUTCOMES:
Any first recurrence (AFR) | 5 years
  defined as any recurrence of ipsilateral chest, breast, regional lymph node recurrence, or distant metastases by Imaging or pathology
Local-regional recurrence free survival (LRFS) | 5 years
  defined as time between randomization and the time of any recurrence of ipsilateral chest, breast, regional lymph node recurrence, distant metastases, or death occurred
Distant metastasis free survival (DMFS) | 5 years
  defined as time between randomization and the time of distant metastases, or death occurred
Recurrence free survival (RFS) | 5 years
  defined as time between randomization and the time of any recurrence of ipsilateral chest, breast, regional lymph node recurrence, distant metastases, or death occurred
Overall Survival (OS) | 5 years
  defined as time between randomization and the time of death occurred
Disease free survival (DFS) | 5 years
  defined as time between randomization and the time of disease recur or death occur
Beast cancer specific mortality (BCSM) | 5 years
  defined as time between randomization and the time of death occur specific due to breast cancer
Patient life quality measurement | 5 years
  At the screening period and after the end of radiotherapy, each group of patients was enrolled in the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Cancer-30 (C30)
Patient life quality measurement | 5 years
  At the screening period and after the end of radiotherapy, each group of patients was enrolled in the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Breast-23 (BR23)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
individual patient data (IPD) will be shared when the research is published.
Supporting Information: Study Protocol
Time Frame: The data will become available in 2030 and forever.
Access Criteria: Study Protocol

REFERENCES:
- [Background] Cheng SH, Horng CF, West M, Huang E, Pittman J, Tsou MH, Dressman H, Chen CM, Tsai SY, Jian JJ, Liu MC, Nevins JR, Huang AT. Genomic prediction of locoregional recurrence after mastectomy in breast cancer. J Clin Oncol. 2006 Oct 1;24(28):4594-602. doi: 10.1200/JCO.2005.02.5676. PMID 17008701
- [Background] Cheng SH, Horng CF, Huang TT, Huang ES, Tsou MH, Shi LS, Yu BL, Chen CM, Huang AT. An Eighteen-Gene Classifier Predicts Locoregional Recurrence in Post-Mastectomy Breast Cancer Patients. EBioMedicine. 2016 Feb 16;5:74-81. doi: 10.1016/j.ebiom.2016.02.022. eCollection 2016 Mar. PMID 27077114
- [Background] Cheng SH, Horng CF, Clarke JL, Tsou MH, Tsai SY, Chen CM, Jian JJ, Liu MC, West M, Huang AT, Prosnitz LR. Prognostic index score and clinical prediction model of local regional recurrence after mastectomy in breast cancer patients. Int J Radiat Oncol Biol Phys. 2006 Apr 1;64(5):1401-9. doi: 10.1016/j.ijrobp.2005.11.015. Epub 2006 Feb 10. PMID 16472935
- [Background] Cheng SH, Tsai SY, Yu BL, Horng CF, Chen CM, Jian JJ, Chu NM, Tsou MH, Liu MC, Huang AT, Prosnitz LR. Validating a prognostic scoring system for postmastectomy locoregional recurrence in breast cancer. Int J Radiat Oncol Biol Phys. 2013 Mar 15;85(4):953-8. doi: 10.1016/j.ijrobp.2012.08.042. Epub 2012 Nov 1. PMID 23122982
- [Background] Cheng SH, Huang TT, Cheng YH, Tan TBK, Horng CF, Wang YA, Brian NS, Shih LS, Yu BL. Validation of the 18-gene classifier as a prognostic biomarker of distant metastasis in breast cancer. PLoS One. 2017 Sep 8;12(9):e0184372. doi: 10.1371/journal.pone.0184372. eCollection 2017. PMID 28886126
- [Background] Huang TT, Pennarun N, Cheng YH, Horng CF, Lei J, Hung-Chun Cheng S. Gene expression profiling in prognosis of distant recurrence in HR-positive and HER2-negative breast cancer patients. Oncotarget. 2018 May 1;9(33):23173-23182. doi: 10.18632/oncotarget.25258. eCollection 2018 May 1. PMID 29796180
- [Background] Pittman J, Huang E, Dressman H, Horng CF, Cheng SH, Tsou MH, Chen CM, Bild A, Iversen ES, Huang AT, Nevins JR, West M. Integrated modeling of clinical and gene expression information for personalized prediction of disease outcomes. Proc Natl Acad Sci U S A. 2004 Jun 1;101(22):8431-6. doi: 10.1073/pnas.0401736101. Epub 2004 May 19. PMID 15152076
- [Background] Huang E, Cheng SH, Dressman H, Pittman J, Tsou MH, Horng CF, Bild A, Iversen ES, Liao M, Chen CM, West M, Nevins JR, Huang AT. Gene expression predictors of breast cancer outcomes. Lancet. 2003 May 10;361(9369):1590-6. doi: 10.1016/S0140-6736(03)13308-9. PMID 12747878
- [Background] Huang TT, Chen AC, Lu TP, Lei L, Cheng SH. Clinical-Genomic Models of Node-Positive Breast Cancer: Training, Testing, and Validation. Int J Radiat Oncol Biol Phys. 2019 Nov 1;105(3):637-648. doi: 10.1016/j.ijrobp.2019.06.2546. Epub 2019 Jul 8. PMID 31295565
- [Derived] Liu J, Tan Y, Bi Z, Huang S, Zhang N, Zhang AD, Zhao L, Wang Y, Liang Z, Hou Y, Xu X, Chen J, Wang F, Lan X, Lin X, Zhang X, Zhou W, Ye X, Guo JG, Wang X, Ding R, Chen J, Huang X. RecurIndex-Guided postoperative radiotherapy with or without Avoidance of Irradiation of regional Nodes in 1-3 node-positive breast cancer (RIGAIN): a study protocol for a multicentre, open-label, randomised controlled prospective, phase III trial. BMJ Open. 2024 Jul 30;14(7):e078049. doi: 10.1136/bmjopen-2023-078049. PMID 39079921